CLINICAL TRIAL: NCT04150913
Title: A Phase 2 Trial of Anakinra for the Prevention of CAR-T Cell Mediated Neurotoxicity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marcela V. Maus, M.D.,Ph.D. (Other)
Collaborators: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor-Investigator, Marcela V. Maus, M.D.,Ph.D., Sponsor-Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-348
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Non Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Relapsed Non Hodgkin Lymphoma; Neurotoxicity; Neurotoxicity Syndromes; Cytokine Release Syndrome
Keywords: Non Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Relapsed Non Hodgkin Lymphoma; Neurotoxicity; Neurotoxicity Syndromes; Cytokine Release Syndrome
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neurotoxicity Syndromes; Cytokine Release Syndrome | interventions — Interleukin 1 Receptor Antagonist Protein; axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Anakinra and Axicabtagene Ciloleucel (Experimental): Patients who meet eligibility criteria for the study will subsequently be enrolled for treatment.
  * Screening
  * Enrollment/Leukapheresis period
  * Bridging therapy (if applicable)
  * Lymphodepleting chemotherapy period
  * Investigational Product (IP) treatment period
    * Anakinra
    * Axicabtagene Ciloleucel
  * Post treatment assessment period
  * Long term follow-up period
  Interventions: Drug: Anakinra; Drug: Axicabtagene Ciloleucel

INTERVENTIONS:
Drug: Anakinra — Subcutaneous, dosage per protocol. Day 0 through Day 6.
  Other Names: Kineret®
Drug: Axicabtagene Ciloleucel — Once, intravenous infusion, dosage per protocol

SUMMARY:
This research study is studying the combination of anakinra and axicabtagene ciloleucel to reduce the occurrence of the side effects Cytokine Release Syndrome (CRS) and neurologic toxicities with relapsed or refractory Non-Hodgkin lymphoma (NHL).

* Relapsed NHL is the condition of returned Non-Hodgkin lymphoma.
* Refractory NHL is the condition of previous treatment resistant Non-Hodgkin lymphoma.
* Cytokine Release Syndrome (CRS) is a group of side effect symptoms that can include nausea, headache, rapid heartbeat, shortness of breath, kidney damage, and rash.
* Neurologic toxicity is nervous system disorder characterized by confusion

This research study involves two drugs:

* Anakinra
* Axicabtagene Ciloleucel.

DETAILED DESCRIPTION:
This Phase 2, single center, open-label research study is studying the combination of Anakinra and Axicabtagene Ciloleucel to reduce the occurrence of the side effects Cytokine Release Syndrome (CRS) and neurologic toxicities in people with relapsed or refractory Non-Hodgkin lymphoma (NHL).

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

* This research study involves two drugs:

  * Anakinra
  * Axicabtagene Ciloleucel
* A total of 20 participants are anticipated to be enrolled to this trial
* The U.S. Food and Drug Administration (FDA) has not approved anakinra for use in treatment of Non-Hodgkin lymphoma (NHL).

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory large B-cell lymphoma after two or more lines of systemic therapy, including diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B-cell lymphoma, high grade B-cell lymphoma, and DLBCL arising from follicular lymphoma.
* At least 1 measurable lesion according to the revised IWG Response Criteria for Malignant Lymphoma 1. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy
* At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis, except for systemic inhibitory/stimulatory immune checkpoint therapy however steroids only require a 7-day washout. At least 3 half-lives must have elapsed from any prior systemic inhibitory/stimulatory immune checkpoint molecule therapy at the time the subject is planned for leukapheresis (e.g. ipilimumab, nivolumab, pembrolizumab, atezolizumab, OX40 agonists, 4-1BB agonists, etc).
* Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for clinically non-significant toxicities such as alopecia)
* Age 18 or older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* ANC ≥1000/uL
* Platelet count ≥75,000/uL
* Absolute lymphocyte count ≥100/uL
* Adequate renal, hepatic, pulmonary and cardiac function defined as:

  * Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min
  * Serum ALT/AST ≤2.5 ULN
  * Total bilirubin ≤1.5 mg/dl, except in subjects with Gilbert's syndrome.
  * Cardiac ejection fraction ≥ 50%, no clinically significant pericardial effusion, and no clinically significant ECG findings
  * No clinically significant pleural effusion
  * Baseline oxygen saturation >92% on room air
* Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential) Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) or follicular lymphoma unless disease free for at least 3 years
* History of Richter's transformation of CLL
* Autologous stem cell transplant within 6 weeks of planned axicabtagene ciloleucel infusion
* History of allogeneic stem cell transplantation
* Prior CD19 targeted therapy with the exception of subjects who received axicabtagene ciloleucel in this study and are eligible for re-treatment
* Prior chimeric antigen receptor therapy or other genetically modified T cell therapy
* History of severe, immediate hypersensitivity reaction attributed to aminoglycosides
* Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management.
* History of HIV infection or acute or chronic active hepatitis B or C infection. Subjects with history of hepatitis infection must have cleared their infection as determined by standard serological and genetic testing per current Infectious Diseases Society of America (IDSA) guidelines.
* Presence of any indwelling line or drain (e.g., percutaneous nephrostomy tube, indwelling Foley catheter, biliary drain, or pleural/peritoneal/pericardial catheter). Dedicated central venous access catheters such as a Port-a-Cath or Hickman catheter are permitted
* Subjects with detectable cerebrospinal fluid malignant cells, or brain metastases, or with a history of CNS lymphoma or primary CNS lymphoma, cerebrospinal fluid malignant cells or brain metastases
* History or presence of CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
* Subjects with cardiac atrial or cardiac ventricular lymphoma involvement
* History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment
* Expected or possible requirement for urgent therapy within 6 weeks due to ongoing or impending oncologic emergency (eg, tumor mass effect, tumor lysis syndrome)
* Primary immunodeficiency
* History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months of enrollment
* Any medical condition likely to interfere with assessment of safety or efficacy of study treatment
* History of severe immediate hypersensitivity reaction to any of the agents used in this study
* Live vaccine ≤ 6 weeks prior to planned start of conditioning regimen
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant. Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential
* Subjects of both genders who are not willing to practice birth control from the time of consent through 6 months after the completion of axicabtagene ciloleucel
* In the investigators judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation
* History of autoimmune disease (e.g. Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt J Frigault, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Frigault MJ, Yao N, Berger TR, Wehrli M, Gallagher KME, Horick N, Graham CE, Jacobson CA, Chen YB, Leick MB, DeFilipp Z, El-Jawahri AR, Johnson PC, Dolaher M, Katsis K, Kim AI, Crombie J, Merryman RW, Cook D, Trailor M, Cho H, Jeffrey R 3rd, Shen R, Filosto S, Nater J, Getz G, Haradhvala NJ, Maus MV. Single-cell dynamics of breakthrough toxicities after anakinra prophylaxis for axicabtagene ciloleucel in lymphoma. Blood Adv. 2025 May 13;9(9):2122-2135. doi: 10.1182/bloodadvances.2024015161. PMID 39928957

RESULTS

PARTICIPANT FLOW:
Groups:
- Anakinra and Axicabtagene Ciloleucel: Patients who meet eligibility criteria for the study will subsequently be enrolled for treatment.
  * Screening
  * Enrollment/Leukapheresis period
  * Bridging therapy (if applicable)
  * Lymphodepleting chemotherapy period
  * Investigational Product (IP) treatment period
    * Anakinra
    * Axicabtagene Ciloleucel
  * Post treatment assessment period
  * Long term follow-up period
  Anakinra: Subcutaneous, dosage per protocol. Day 0 through Day 13.
  Axicabtagene Ciloleucel: Once, intravenous infusion, dosage per protocol
Period: Overall Study
Arm/Group | Anakinra and Axicabtagene Ciloleucel
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Anakinra and Axicabtagene Ciloleucel
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 2
  Unknown or Not Reported | 2
International Prognostic Index [Median (Full Range); unit: Score (0-5)] — The IPI is a score used to predict how aggressive a person's non-Hodgkin lymphoma might be. It is based on five things measured before treatment: Age over 60, High levels of a blood enzyme called LDH, Trouble with daily activities (performance status), Cancer in many lymph nodes or areas (stage III or IV), Cancer outside the lymph nodes in more than one place.
  Each item adds 1 point to the total score.
  Score Range: 0 to 5
  What the Scores Mean: A lower score (0-1) means a better outlook; A higher score (4-5) means a more serious outlook
  When It's Measured: Before treatment starts
  Score (0-5) | 3 [0 to 4]
Eastern Cooperative Oncology Group [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale used to assess a patient's level of functioning. It ranges from 0 (fully active) to 5 (dead), with lower scores indicating better performance status.
  Participants
    Grade 0 | 5
    Grade 1 | 10
Histology [Count of Participants; unit: Participants]
  tFL | 5
  DLBCL NOS | 9
  HGBCL | 1
Number of prior regimens [Count of Participants; unit: Participants]
  Primary refractory disease | 3
  Prior autologous HSCT | 3
Tumor burden, Baseline LDH (U/L) [Median (Full Range); unit: U/L] | 223 [165 to 2022]
Tumor burden, Baseline SPD (mm2) [Median (Full Range); unit: mm2] | 2239 [542 to 13807]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Neurotoxicity as Per CTCAE v4.03 Criteria
Description: The incidence of grade 2+ neurotoxicity is reported below and was assessed using CTCAE (Common Terminology Criteria for Adverse Events) v4.04 criteria. Neurotoxicity is a serious side effect of cancer treatments that can impact the central and peripheral nervous systems. Neurotoxicity manifestations vary and can include confusion, obtundation, seizures, hallucinations, aphasia, ataxia, and more rarely, profound cerebral edema.
Time Frame: 30 Days
Population: Neurotoxicity, Max Grade
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra and Axicabtagene Ciloleucel
Number analyzed (Participants) | 15
Participants
  Grade 1 | 3
  Grade 2 | 2
  Grade 3-4 | 5
  Grade 5 | 1
  Did not experience Neurotoxicity | 4

2. Secondary Outcome: Objective Response Rate
Description: Objective response rate (ORR) is defined as the incidence of either a complete response (CR) or a partial response (PR) by the revised IWG Response Criteria for Malignant Lymphoma. All participants who don't meet the ORR criteria by the analysis data cutoff date will be considered non-responders.
  * CR = complete disappearance of all detectable clinical evidence of disease and disease related symptoms if present before therapy; PET scan negative; lymph nodes/nodal masses regressed to normal size; normal size spleen/liver on CT scan; bone marrow aspirate and biopsy shows no evidence of disease by morphology or negative by IHC.
  * PR = ≥ 50% decrease in sum of the product of diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses; no size increase of nodes/liver/spleen; no new sites of disease; post-treatment PET scan positive in ≥ 1 previously involved site.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra and Axicabtagene Ciloleucel
Number analyzed (Participants) | 15
Participants
  Overall Response Rate | 13
  Complete Response | 7
  Partial Response | 6

3. Secondary Outcome: Duration of Response
Description: Among participants who experience an objective response, duration of response (DOR) is defined as the date of their first objective response to disease progression per the revised IWG Response Criteria for Malignant Lymphoma, or death regardless of cause. Participants not meeting the criteria for progressive disease (PD) or death by the analysis data cutoff date will be censored at their last evaluable disease assessment date and their response will be noted as ongoing.
  * PD = ≥ 50% increase from nadir in the sum of the products of at least two lymph nodes; ≥ 50% increase in product of the diameters of single node; new lesion >1.5 cm; ≥ 50% size increase of splenic/hepatic nodules; ≥ 50% increase in longest diameter of any single previously identified node more than 1 cm in its short axis; PET scan positive
Time Frame: first objective response to disease progression death regardless of cause up 24 Months
Population: Progression Free Survival (PFS); Overall Survival OS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Anakinra and Axicabtagene Ciloleucel: Patients who meet eligibility criteria for the study will subsequently be enrolled for treatment.
  * Screening
  * Enrollment/Leukapheresis period
  * Bridging therapy (if applicable)
  * Lymphodepleting chemotherapy period
  * Investigational Product (IP) treatment period
    * Anakinra
    * Axicabtagene Ciloleucel
  * Post treatment assessment period
  * Long term follow-up period
  Anakinra: Subcutaneous, dosage per protocol. Day 0 through Day 6.
  Axicabtagene Ciloleucel: Once, intravenous infusion, dosage per protocol
Arm/Group | Anakinra and Axicabtagene Ciloleucel
Number analyzed (Participants) | 15
percentage of participants
  PFS at 6 months | 58.2 [29.4 to 78.7]
  PFS at 12 months | 42.4 [16.9 to 66.1]
  OS at 6 months | 79.4 [48.8 to 92.9]
  OS at 12 months | 64.2 [33.9 to 83.4]

4. Secondary Outcome: Progression-free Survival
Description: Kaplan-Meier estimates and 2-sided 95% confidence intervals will be generated for progression-free survival time
Time Frame: infusion date to the date of disease progression or death from any cause up 24 Months
Population: Progression Free Survival
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anakinra and Axicabtagene Ciloleucel
Number analyzed (Participants) | 15
percentage of participants
  PFS at 6 months | 58.2 [29.4 to 78.7]
  PFS at 12 months | 42.4 [16.9 to 66.1]

5. Secondary Outcome: Overall Survival
Description: Kaplan-Meier estimates and 2-sided 95% confidence intervals will be generated for OS.
Time Frame: time from axicabtagene ciloleucel infusion to the date of death or analysis data cutoff date will be censored at last contact date up to 24 months.
Population: Overall Survival
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anakinra and Axicabtagene Ciloleucel
Number analyzed (Participants) | 15
percentage of participants
  OS at 6 months | 79.4 [48.8 to 92.9]
  OS at 12 months | 64.2 [33.9 to 83.4]

6. Secondary Outcome: Number of Participants With Adverse Events CTCAE Version 4.03 Grade 3 or Higher
Description: Subject incidence rates of adverse events including all, serious, fatal, CTCAE version 4.03 Grade 3 or higher and treatment related AEs reported throughout the conduct of the study will be tabulated by preferred term and system organ class
Time Frame: 24 Months
Population: Participants who experienced Adverse Events (AE), Grade 3 or higher
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra and Axicabtagene Ciloleucel
Number analyzed (Participants) | 15
Participants
  Infections and Infestations: Grade 3 | 4
  Infections and Infestations : Grade 4 | 1
  Infections and Infestations : Grade 5 | 1
  Nervous System Disorders : Grade 3 | 6
  Nervous System Disorders : Grade 4 | 1
  Blood and lymphatic system disorders : Grade 3 | 9
  Blood and lymphatic system disorders : Grade 4 | 1
  Cardiac disorders : Grade 3 | 1
  Ear and labyrinth disorders : Grade 3 | 1
  Endocrine disorders : Grade 3 | 1
  Endocrine disorders : Grade 4 | 1
  Gastrointestinal disorders : Grade 3 | 4
  General disorders and administration site conditions : Grade 3 | 5
  Hepatobiliary disorders : Grade 3 | 1
  Immune system disorders : Grade 3 | 1
  Investigations : Grade 3 | 9
  Investigations : Grade 4 | 9
  Metabolism and nutrition disorders : Grade 3 | 9
  Metabolism and nutrition disorders : Grade 4 | 1
  Musculoskeletal and connective tissue disorders : Grade 3 | 2
  Psychiatric disorders : Grade 3 | 2
  Renal and urinary disorders : Grade 3 | 2
  Respiratory, thoracic and mediastinal disorders : Grade 3 | 5
  Vascular disorders : Grade 3 | 4
  Vascular disorders : Grade 4 | 1

7. Secondary Outcome: Rate of Cytokine Release Syndrome (CRS) as Per Lee 2014 for CRS
Description: The incidence of max grade 2+ CRS will be assessed
Time Frame: Within 30 days after infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Anakinra and Axicabtagene Ciloleucel
Number analyzed (Participants) | 15
Participants
  Grade 2 | 6
  Grade 3 | 1
  Grade 4 | 1
  Grade 1 | 6
  No CRS | 1

ADVERSE EVENTS:
Time Frame: All adverse events observed by the investigator or reported by the subject that occur from enrollment through 3 months were monitored and reported. After 3 months, only targeted adverse events including (eg, neurological, hematological, infections, autoimmune disorders, and secondary malignancies) were monitored and reported for 24 months.
Arm/Group | Anakinra and Axicabtagene Ciloleucel
All-Cause Mortality (participants affected / at risk) | 7/15
Serious Adverse Events (participants affected / at risk) | 9/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra and Axicabtagene Ciloleucel (N=15)
Upper Respiratory Infection (Infections and infestations) | 2 (2)
Hypotension (Vascular disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Vasovagal Reaction (Nervous system disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Immune effector cell-associated neurotoxicity syndrome (ICANS) (Nervous system disorders) | 2 (3)
Cytokine Release Syndrome (CRS) (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra and Axicabtagene Ciloleucel (N=15)
Abdominal pain (Gastrointestinal disorders) | 6 (10)
Bloating (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 9 (11)
Dry Mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (3)
Fecal incontinence (Gastrointestinal disorders) | 3 (3)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 11 (16)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (7)
Ulcerative Colitis (Gastrointestinal disorders) | 1 (1)
Hemoptysis/Melena (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (13)
Anemia (Blood and lymphatic system disorders) | 11 (41)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (3)
Tachycardia-Bradycardia Syndrome (Cardiac disorders) | 1 (1)
Pulmonary Embolism (Cardiac disorders) | 1 (1)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 2 (3)
Sinus Tachycardia (Cardiac disorders) | 2 (7)
Ventricular Tachycardia (Cardiac disorders) | 2 (2)
Hearing Impaired (Ear and labyrinth disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Adrenal Insufficiency (Endocrine disorders) | 1 (4)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Eye Irritation (Eye disorders) | 1 (1)
Right Conjunctival Hemorrhage (Eye disorders) | 1 (1)
Periorbital Edema (Eye disorders) | 1 (1)
Vision Decreased (Eye disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Edema Limbs (General disorders) | 2 (3)
Fatigue (General disorders) | 15 (23)
Fever (General disorders) | 7 (18)
Flu like symptoms (General disorders) | 1 (1)
Gait Disturbance (General disorders) | 1 (1)
Generalized Edema (General disorders) | 4 (5)
Injection Site Reaction (General disorders) | 1 (1)
Localized Edema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Hickman Line Irritation (General disorders) | 1 (1)
Central Line Irritation (General disorders) | 1 (1)
Distributive Shock (General disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Gallbladder Obstruction (Hepatobiliary disorders) | 1 (1)
Portal Vein Thrombosis (Hepatobiliary disorders) | 1 (2)
Cytokine Release Syndrome (Immune system disorders) | 14 (22)
Seasonal Allergies (Immune system disorders) | 2 (2)
Systemic Inflammatory Response Syndrome (Immune system disorders) | 1 (1)
Hypogammaglobulinemia (Immune system disorders) | 2 (2)
Bacteremia (Infections and infestations) | 1 (1)
Enterocolitis Infectious (Infections and infestations) | 2 (2)
COVID Infection (Infections and infestations) | 2 (3)
Otitis Media (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 2 (2)
Thrush (Infections and infestations) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 2 (5)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Activated Partial Thromboplastin Time-Prolonged (Investigations) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 5 (5)
Alkaline Phosphatase Increased (Investigations) | 4 (4)
Aspartate Aminotransferase Increased (Investigations) | 4 (4)
Blood Bilirubin Increased (Investigations) | 1 (3)
Creatinine Increased (Investigations) | 1 (2)
Fibrinogen Decreased (Investigations) | 1 (1)
Lipase Increased (Investigations) | 1 (1)
Hypogammaglobulinemia (Investigations) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 7 (37)
Neutrophil Count Decreased (Investigations) | 9 (40)
Platelet Count Decreased (Investigations) | 8 (24)
Serum Amylase Increased (Investigations) | 1 (1)
Weight Loss (Investigations) | 1 (1)
White Blood Cell Decreased (Investigations) | 1 (10)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 11 (20)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (6)
Hyperlipidemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (9)
Hypokalemia (Metabolism and nutrition disorders) | 3 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (10)
Hyponatremia (Metabolism and nutrition disorders) | 4 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (8)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized Upper Body Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Intermittent Jaw Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed Level of Consciousness (Nervous system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 7 (9)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (2)
Edema Cerebral (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 3 (5)
Headache (Nervous system disorders) | 10 (17)
Memory Impairment (Nervous system disorders) | 1 (1)
Muscle Weakness Right-Sided (Nervous system disorders) | 1 (1)
Olfactory Nerve Disorder (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral Motor Neuropathy (Nervous system disorders) | 4 (4)
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (2)
Tremor (Nervous system disorders) | 5 (8)
Vasovagal Reaction (Nervous system disorders) | 1 (1)
Hyperalgesia (Nervous system disorders) | 1 (3)
Aphasia (Nervous system disorders) | 1 (3)
Altered Mental Status (Nervous system disorders) | 1 (4)
Word Finding Difficulties (Nervous system disorders) | 1 (1)
Peripheral Neuropathy (Nervous system disorders) | 1 (1)
Intermittent Delayed Word (Nervous system disorders) | 1 (1)
Emotional Lability (Nervous system disorders) | 1 (1)
Expressive Aphasia (Nervous system disorders) | 1 (1)
Subarachnoid Hemorrhage (Nervous system disorders) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1)
Neurotoxicity (Nervous system disorders) | 2 (3)
Agitation (Psychiatric disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 5 (5)
Confusion (Psychiatric disorders) | 5 (12)
Delirium (Psychiatric disorders) | 3 (4)
Depression (Psychiatric disorders) | 2 (2)
Hallucinations (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (7)
Acute Kidney Injury (Renal and urinary disorders) | 3 (4)
Dysuria (Renal and urinary disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 2 (2)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
Secondary Infertility (Reproductive system and breast disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulceration (Skin and subcutaneous tissue disorders) | 3 (3)
Leg Petechia (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 6 (18)
Thromboembolic Event (Vascular disorders) | 1 (1)
Right Upper Extremity DVT (Vascular disorders) | 1 (1)
Right Lower Extremity Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Immune effector cell-associated neurotoxicity syndrome (ICANS) (Nervous system disorders) | 10 (32)

LIMITATIONS AND CAVEATS:
Limited number of patients enrolled into the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT04150913/Prot_SAP_000.pdf